CLINICAL TRIAL: NCT02684513
Title: Impact of Oral Carbohydrate Consumption Prior to Cesarean Section on Preoperative Well-being
Brief Title: Impact of Oral Carbohydrate Consumption Prior to Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Heermann Anesthesia Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB201501150
Record Dates: First submitted 2016-02-04; First posted 2016-02-18 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Dehydration
Keywords: Well-being; Quality of Recovery; Maternal complications
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral Carbohydrate Beverage Group (Active Comparator): Subjects assigned to this group will receive 710 mL of a preoperative beverage the evening prior to surgery and 355 mL the morning of surgery.
  Interventions: Dietary Supplement: Oral Carbohydrate Beverage
- Rehydration Beverage Group (Active Comparator): Subjects assigned to this group will receive 710 mL of re-hydration beverage the evening prior to surgery and 355 mL the morning of surgery.
  Interventions: Dietary Supplement: Rehydration beverage
- Fasted Controls (No Intervention): Subjects assigned to this group will fast for ≥8 hours prior to surgery.

INTERVENTIONS:
Dietary Supplement: Oral Carbohydrate Beverage — The oral carbohydrate beverage will be consume in a 710 mL amount the evening prior to surgery and then a 355 mL amount the morning of surgery.
  Other Names: Preoperative beverage
  Arms: Oral Carbohydrate Beverage Group
Dietary Supplement: Rehydration beverage — The rehydration beverage group will be consume in a 710 mL amount the evening prior to surgery and then a 355 mL amount the morning of surgery.
  Other Names: Preoperative beverage
  Arms: Rehydration Beverage Group

SUMMARY:
For more than 15 years, traditional fasting regimens prior to scheduled surgeries have been called into question, yet prolonged preoperative fasting remains common practice. While prolonged fasting is aimed at reducing the risk of pulmonary aspiration, prolonged fasting is uncomfortable, has an inconsistent effect on gastric volumes and acidity and may lead to dehydration without a clear reduction in the incidence of aspiration. Fasting by itself decreases hepatic glycogen stores, induces a state of insulin resistance and impairs cardiovascular function. Yet, prolonged preoperative fasting remains common.

Preoperative oral carbohydrate (CHO) consumption improves insulin sensitivity and decreases the time to return of gut function without increasing gastric volumes or acidity compared to other clear liquids and fasting. Previous work has shown oral CHO consumption improves patient well-being to a greater degree than placebo drink (water or flavored water) and fasted controls. Oral CHO also outperforms a similar volume of intravenous glucose supplementation. These benefits have reduced hospital stays in a variety of surgical models by as much as 20%. Further, preoperative CHO supplementation improved postoperative patient hunger, thirst, anxiety, fatigue and nausea.

The purpose of this research study is to determine if drinking a high carbohydrate beverage before cesarean section surgery can improve patient well-being, compared to patients who drink a low carbohydrate beverage or fast before surgery.

DETAILED DESCRIPTION:
The study hopes to determine if either of two different oral beverages (a higher CHO concentration versus a lower CHO concentration) is superior to routine fasting in terms of preoperative well-being among patients presenting for scheduled cesarean section. Preoperative well-being will be determined by a composite of visual analog scale scores aimed at assessing hunger, thirst, anxiety, fatigue and nausea on the morning of surgery.

Women will be recruited from one of two outpatient obstetric clinics, University of Florida (UF) Health Women's Center - Medical Plaza or UF Health Women's Center. Women presenting for scheduled cesarean section will be provided with an opportunity to participate. Then the women will be randomized into one of three groups: oral carbohydrate beverage (group CHO), re-hydration beverage of an equal volume (group R) or fasted controls (group F). All subjects who consent to participation will have the following recorded: height, weight, age, indication for cesarean section, surgeon, and number of prior cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* Full-term (≥37 weeks gestation) with singleton gestation
* Proficient with English language
* Planning on undergoing scheduled cesarean delivery under neuraxial anesthesia

Exclusion Criteria:

* Women with pre-gestational or gestational diabetes mellitus or diabetes present prior to pregnancy
* Women who did not complete a gestational diabetes screening test
* Women who received steroids within the past 7 days prior to delivery
* Women who received magnesium sulfate in the setting of hypertensive disorders of pregnancy
* Women with a history of chronic opioid use
* Preterm pregnancies
* Fetuses with congenital abnormalities or growth restriction
* Multiple gestation
* Women who are American Society of Anesthesiology Class III or higher

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Change in preoperative well-being assessment from baseline to one hour using the 100 millimeter (mm) visual analogue scale. | Change from baseline to one hour
  100 mm visual analogue scales for hunger, thirst, anxiety, fatigue and nausea administered on the morning of surgery prior to morning beverage consumption and 60 minutes after the beverage. All measurements will be assessed using the same scale starting at 0 to 100mm with 0 being the worst and 100 being the best and average being 85.

SECONDARY OUTCOMES:
Changes between the maternal groups assessed by the mean arterial pressure (MAP) recordings in every 5 minute period | At time of surgery to the conclusion
  Maternal cardiovascular function will be assessed by using the average of all the mean arterial pressure (MAP) recordings in every 5 minute period. This will be measured by using a student's t-test for significant differences between the groups.
Number of participants admitted to maternal intensive care unit between the groups | Up to 15 days
  Number of ICU admissions during hospitalization between the groups
Number of days in the hospital for each participant between the groups | Up to 15 days
  Number of days in the hospital for each participant between the groups. This will be measured by using the chi-square tests to assess the frequency of this outcome between the groups.
Number of postoperative infections between the groups | Up to 15 days
  Number of postoperative infections for each participant between the groups. This will be measured by using the chi-square tests to assess the frequency of this outcome between the groups.
Neonates with plasma glucose level of less than 45 mg/dL between the groups | Baseline
  First umbilical cord blood sample will be taken for plasma glucose level of less than 45 mg/dL to note hypoglycemia between the groups.
Number of neonates with a 5 minute Apgar score less than 7 between the groups | 5 minutes
  Record of the 5 minute apgar score < 7. Apgar scores are as follows: between 7 and 10, means the neonate is in good shape, between 4 and 6 may need some help breathing, and 3 or less may need immediate lifesaving measures.
Number of neonates on ventilation for 6 hours or greater between the groups | 6 hours
  Number of neonates on ventilation for 6 hours or greater will be recorded.
Number of neonates diagnosed with an infection between the groups. | Baseline
  Number of neonates with an infection diagnosis. This will be measured by using the chi-square tests to assess the frequency of this outcome between the groups.
Number of neonates admitted to the intensive care unit (ICU) between the groups | Baseline
  Number of neonates admitted to the ICU between the groups. This will be measured by using the chi-square tests to assess the frequency of this outcome between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wendling, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wendling AL, Byun SY, Koenig M, Vasilopoulos T. Impact of oral carbohydrate consumption prior to cesarean delivery on preoperative well-being: a randomized interventional study. Arch Gynecol Obstet. 2020 Jan;301(1):179-187. doi: 10.1007/s00404-020-05455-z. Epub 2020 Feb 5. PMID 32025843